CLINICAL TRIAL: NCT06305910
Title: Phase I Trial: CD200 Activation Receptor Ligand (CD200AR-L) and Allogeneic Tumor Lysate Vaccine Immunotherapy With Adjuvant Reirradiation for Recurrent High-Grade Glioma and Newly Diagnosed Diffuse Midline Glioma/Diffuse Intrinsic Pontine Glioma in Children and Young Adults
Brief Title: CD200AR-L and Allogeneic Tumor Lysate Vaccine Immunotherapy for Recurrent HGG and Newly Diagnosed DMG/DIPG in Children and Young Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OX2 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CMN-DMGVac-01
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Diffuse Midline Glioma, H3 K27M-Mutant; Recurrent High Grade Glioma
MeSH Terms: conditions — Glioma | interventions — Therapeutics; Imiquimod; Radiation

STUDY DESIGN:
Intervention Model Description: 3+3 design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CD200AR-L (Experimental): Up to 3 dose levels (2.0, 3.75, and 5.0 micrograms/kg/dose) of CD200AR-L will be tested with a Dose Level -1 (1.0 microgram/kg/dose) in the event of toxicity at the 2.0 micrograms/kg/dose level. This will be given with fixed doses of 1mg GBM6-AD vaccine and topical imiquimod. A single dose of 300cGy re-irradiation will be given on Day 15. Patients with DMG/DIPG must have completed standard-of-care radiation before enrolling.
  The MTD will be identified using the standard 3+3 design. Upon determination of the MTD, additional patients will be enrolled as part of an expansion cohort. This study will first enroll patients ≥ 12 years of age into Dose Level 1 in order to acquire safety data prior to subsequent enrollment of study subjects aged 2-11 years.
  Interventions: Drug: Treatment with CD200AR-L

INTERVENTIONS:
Drug: Treatment with CD200AR-L — Treatment with CD200AR-L (up to 3 dose levels of CD200AR-L with a Dose Level -1 in the event of toxicity) with fixed doses of GBM6-AD vaccine. Each patient will also be given topical imiquimod and a single dose of 300cGy re-irradiation.
  Other Names: Imiquimod; GBM6-AD; Single dose of radiation (300 cGy)

SUMMARY:
This is a single center Phase I study of a new adjuvant CD200 activation receptor ligand, CD200AR-L, in combination with imiquimod and GBM6-AD vaccine to treat malignant glioma in children and young adults.

The primary objective of this study is to determine the maximum tolerated dose (MTD) of CD200AR-L when given with a fixed dose of GBM6-AD vaccine, imiquimod, and a single dose of radiation for patients with recurrent High Grade Glioma (HGG) or following standard of care therapy radiation therapy for newly diagnosed Newly Diagnosed Diffuse Midline Glioma/Diffuse Intrinsic Pontine Glioma (DIPG/DMG).

DETAILED DESCRIPTION:
A previous pediatric trial using GBM6-AD vaccine was found to be safe, and an appropriate pediatric dose of GBM6-AD was determined, but the efficacy of the vaccine was diminished due to secretion of CD200 by the patient's HGG or DMG/DIPG cells. CD200 is known to binds to CD200 inhibitory receptor (CD200R1) on immune cells and suppress the immune cell response. Laboratory studies have shown that administering agents that bind to the CD200 activation receptor (CD200-AR) on immune cells results in activation of immune cells and overcomes any inhibitory signals caused by CD200.

CD200AR-L is a newly developed agent that binds to CD200-AR. This trial will assess the combination of CD200AR-L with GBM6-AD vaccine, imiquimod cream and a single dose of radiation given on day 15 for the treatment of recurrent HGG and newly diagnosed DMG/DIPG.

This study has the following primary goals:

1. To determine the maximum tolerated dose and side-effects of the experimental medicine, CD200AR-L, when given with a fixed dose of GBM6-AD vaccine in combination with imiquimod cream and a single dose of radiation on Day 15 for patients with recurrent HGG or newly diagnosed DMG/DIPG in children.
2. To use the information from this study to design a larger study of the GBM6-AD vaccine and CD200AR-L treatment to assess the effectiveness of this combination vaccine in pediatric HGG and newly diagnosed DMG/DIPG.

Study treatment consists of CD200AR-L, GBM6-AD vaccine and imiquimod, along with a single dose of radiation on day 15. Study treatment will begin approximately 14 days after the completion of standard of care radiation therapy for patients with newly diagnosed DMG/DIPG and at the time of recurrence for patients with HGG. The study will enroll patients between the ages of 2 - 25 years, but it will initially enroll and treat 3 patients age > 12 years in the first dosing cohort in order to acquire safety data before enrolling patients 2-11 years of age. Up to 3 dose levels of CD200AR-L will be tested, with dose reduction in the event of toxicity.

Each vaccine treatment is given as an outpatient visit on two consecutive days. Imiquimod cream is applied to the supraclavicular site followed by 2 supraclavicular injections of CD200AR-L each day for 2 consecutive days. On the second day, following application of Imiquimod cream and CD200AR-L injection, 2 supraclavicular injections of GBM6-AD vaccine will be given. All CD200AR-L and GBM6-AD vaccine administrations must be done at Children's Minnesota. Two-day injection series will be administered every week for the first 3 weeks, then every 4 weeks starting at week 7 for the next 8 weeks, then every 8 weeks starting at week 19 for 2 years. On day 15, a single dose of 300 cGy radiation will be given to help sensitize the tumor to immune attack. The patient will undergo a series of MRIs to follow the status of their tumor, blood work for immune characterization, and pediatric functional performance assessments. Treatment will continue for 2 years, unless disease progression is noted on MRI, unacceptable toxicity develops, a greater than 8-week treatment delay occurs during the maintenance phase, or the patient withdraws from the study. The patient will have an option of continuing therapy beyond 2 years if they are tolerating the treatment and if their tumor is controlled by the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed DIPG/DMG with documented H3K27M alteration (based on IHC or DNA sequencing performed in a CLIA-certified laboratory) or recurrent HGG. Patients cannot enroll until they are a minimum of 14 days and preferably within 30 days from the last dose of radiation.
* Diagnosis of recurrent HGG based on MRI findings. Recurrent HGG must have received standard of care radiation at diagnosis. Prior biopsy material will be required to confirm diagnosis of HGG; however, biopsy of the recurrent/progressive lesion will not be required for study enrollment.
* Maximal safe resection is preferred prior to clinical trial enrollment if indicated and feasible.
* Clinically stable on a dose of corticosteroids not to exceed an equivalent of dexamethasone 0.1 mg/kg/day (maximum 4 mg) for at least 2 weeks prior to study enrollment.
* Prior therapy wash-out is required
* Minimum of 28 days since last dose of any targeted therapy (including bevacizumab), immunotherapy, investigational agents.
* Minimum of 10 days since any anti-cancer intervention: cytoreductive surgery/laser ablation and a minimum of 28 days since any viral therapy
* Voluntary written consent obtained by patient if ≥18 years of age or a parent or guardian if <18 years of age before the performance of any study-related procedure not part of standard medical care
* Able to comply with follow-up visit schedule (i.e., return to clinic for follow-up visits).
* Willing to allow for collection of pre-treatment research related blood collection [1-5 mL red top tube and 2-10 mL green top tubes (or to a max of 2 ml/kg of body weight)] for immune characterization. If a patient does not subsequently enroll in the study, the samples will be destroyed according to institutional protocol.
* Lansky play performance score ≥60 (<16 years) or Karnofsky (≥16 years) performance score of ≥60
* Sexually active persons of child-bearing potential or with partners of childbearing potential must agree to use a highly effective form of contraception during the 2-year treatment period. Urine pregnancy tests will be obtained at defined time points during protocol therapy.
* Adequate bone marrow reserve: Absolute neutrophil (segmented and bands) count (ANC) ≥1.0 x 10E9/L, platelets ≥75 x 10E9/L; Hemoglobin ≥8 g/dL
* Hepatic: Bilirubin ≤1.3 mg/dL and SGPT (ALT) ≤2.5 x upper limit of normal (ULN) for age
* Renal: Normal serum creatinine for age or creatinine clearance >60 ml/min/1.73 mE2

Exclusion Criteria:

* Known sensitivity to the GBM6-AD tumor lysate vaccine, CD200AR-L, or imiquimod.
* Unable to complete a standard upfront course of radiotherapy due to disease progression or intolerance of therapy.
* Radiographic evidence of diffuse leptomeningeal disease.
* Prior history of malignancy within 5 years of enrollment.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
* Concurrent use of tumor treatment field devices (e.g., Optune) - permitted until the time of consent.
* History of any laboratory findings consistent with any uncontrolled immune system abnormalities such as hyper-immunity (e.g., autoimmune diseases, thyroid dysfunction, lupus, scleroderma, etc.) and hypo-immunity [e.g., myelodysplastic disorders, marrow failures, human immunodeficiency virus/acquired immunodeficiency syndrome (HIV/AIDS), transplant immune-suppression, etc.]. Any known autoimmune disease must be clinically silent and without associated laboratory abnormalities for at least 1 year in the absence of any disease directed therapy or systemic steroids.
* Any conditions that could potentially alter immune function (e.g., HIV/AIDS, hepatitis B, untreated hepatitis C, multiple sclerosis, renal failure).
* Receiving ongoing treatment with any immunosuppressive drug for any reason, excluding those patients requiring a low dose of corticosteroids equivalent to dexamethasone 0.1 mg/kg/day (maximum 4 mg) or less for treatment of tumor-related edema.
* Not able to tolerate an MRI or radiation therapy even with reasonable accommodations or sedation.
* Known pregnancy or anticipated conception during the 1-year study period

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of CD200AR-L | 24 months
  Maximum tolerated dose (MTD) of CD200AR-L when administered with imiquimod and GBM6-AD vaccine to treat High-Grade Glioma (HGG) and Newly Diagnosed Diffuse Midline Glioma/Diffuse Intrinsic Pontine Glioma (DMG/DIPG) in children and young adults.

SECONDARY OUTCOMES:
Incidence of serious adverse events (SAEs) | 24 months
Time to progression (TTP) by 24 months | 24 months
Progression free survival (PFS) by 24 months | 24 months
Overall survival (OS) by 24 months | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Minnesota, Minneapolis, Minnesota, United States